CLINICAL TRIAL: NCT06443606
Title: Efficacy and Safety of Bezafibrate 400 mg and Bezafibrate 200 mg as Adjunctive Treatments in Patients With Primary Biliary Cholangitis and Non-optimal Biochemical Response to Ursodeoxycholic Acid Therapy: a 12-month, Double-blind, Randomized, Placebo-controlled Trial With a 12-month, Double-blind, Placebo-free Extension Phase.
Brief Title: Efficacy and Safety of Bezafibrate 400 mg and Bezafibrate 200 mg as Adjunctive Treatments in Patients With Primary Biliary Cholangitis and Non-optimal Biochemical Response to Ursodeoxycholic Acid Therapy
Acronym: BEZURSO 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP220822
Record Dates: First submitted 2024-02-21; First posted 2024-06-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: BPC; Non Optimal Response to UDCA
Keywords: Bezafibrate; PBC; Digestive System Diseases; Ursodeoxycholic Acid
MeSH Terms: conditions — Digestive System Diseases | interventions — Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bezafibrate 400 mg group in addition to UDCA therapy (Experimental): Bezafibrate 400 mg and Placebo of Bezafibrate 200 mg until 48 weeks in double blind
  Interventions: Drug: Bezafibrate 400 mg in addition to UDCA therapy
- Bezafibrate 200 mg group in addition to UDCA therapy (Experimental): Bezafibrate 200 mg and Placebo of Bezafibrate 400 mg until 96 weeks in double blind.
  Interventions: Drug: Bezafibrate 200 mg in addition to UDCA therapy
- Placebo group in addition to UDCA therapy (Placebo Comparator): Placebo of Bezafibrate 400 mg Placebo of Bezafibrate 200 mg until 48 weeks in double blind. And follow-up extension phase of bezafibrate 400 mg and bezafibrate 200 mg until 48 weeks in double blind.
  Interventions: Drug: Placebo in addition to UDCA therapy

INTERVENTIONS:
Drug: Bezafibrate 400 mg in addition to UDCA therapy — * Bezafibrate 400 mg and Placebo of Bezafibrate 200 mg in addition to continued UDCA at minimum dose of 12 mg/kg/d.
  * Duration 96 weeks bezfibrate/ UDCA = daily oral dose.
  Arms: Bezafibrate 400 mg group in addition to UDCA therapy
Drug: Bezafibrate 200 mg in addition to UDCA therapy — * Bezafibrate 200 mg and Placebo of Bezafibrate 400 mg in addition to continued UDCA at minimum dose of 12 mg/kg/d.
  * Duration 96 weeks bezfibrate/ UDCA = daily oral dose.
  Arms: Bezafibrate 200 mg group in addition to UDCA therapy
Drug: Placebo in addition to UDCA therapy — * Placebo of Bezafibrate 400 mg and Placebo of Bezafibrate 200 mg in addition to continued UDCA at minimum dose of 12 mg/kg/d.
  * Duration 96 weeks placebo /UDCA = daily oral dose.
  Arms: Placebo group in addition to UDCA therapy

SUMMARY:
Primary biliary cholangitis (PBC) is a rare chronic, progressive, cholestatic liver disease that leads to cirrhosis and its life-threatening complications if undertreated. Ursodeoxycholic acid (UDCA) is the standard-of-care therapy for PBC. However, patients with an inadequate biochemical response to UDCA according to the Paris-2 criteria are still at high-risk of poor clinical outcome. In this situation of biochemical resistance to UDCA, bezafibrate 400 mg/d given in association with UDCA has been shown to improve the symptoms, biochemical response (BEZURSO study), histologic features, and possibly long-term clinical outcome. However, it has been shown that even patients with an adequate response to UDCA but persistent elevation in biochemical markers of cholestasis or liver inflammation, including alkaline phosphatases (ALP), gamma-glutamyl transpeptidase (GGT), transaminases, or total bilirubin (i.e., non-optimal biochemical response) have still an increased risk of death or liver transplantation in the long term, thus defining the complete normalization of these markers as the new clinically-relevant target for PBC treatment. In parallel to these findings, bezafibrate 400 mg/d as a second-line therapy for PBC could be associated with potentially dose-related, muscle, kidney, or liver toxic effects, and whether bezafibrate 200 mg/d could have a better benefit/risk ratio in this disease-setting remains to be determined. Therefore, our aim is to evaluate the efficacy and safety of bezafibrate 400 mg and bezafibrate 200 mg as adjunctive treatments in PBC patients with non-optimal biochemical response to UDCA.

DETAILED DESCRIPTION:
The study is a phase-3 multicenter, randomized, parallel-group (1:1:1), placebo-controlled trial with a 12-month, double-blind, placebo-free extension phase.

It evaluates the efficacy and safety of bezafibrate 400 mg and bezafibrate 200 mg as adjunctive treatments in patients with PBC with an non-optimal biochemical response to UDCA.

Treatments groups :

Arm 1: Bezafibrate 400 mg and Placebo of Bezafibrate 200 mg until 96 weeks in double blind.

Arm 2: Bezafibrate 200 mg and Placebo of Bezafibrate 400 mg until 96 weeks in double blind.

Arm 3: Placebo of Bezafibrate 400 mg and Placebo of Bezafibrate 200 mg until 48 weeks in double blind. Then follow-up extension phase of bezafibrate 400 mg or bezafibrate 200 mg (second randomization) until 48 weeks in double blind.

Assessement: Study visits at Inclusion, Randomisation (M0) and then every 3 months until W48 and extension until W96. In accordance with routine care, an additional follow-up is added between 108 and 120 weeks

32 sites within the French network of reference and competence centres for rare liver diseases FILFOIE will participate.

No interim analysis planned. Analysis will be performed at the end of the study after data reviewed and data base locked according to the intent to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 80 years
* Diagnosis of PBC based on at least 2 of the following criteria (EASL clinical practice guidelines 2017):

  * Elevated ALP level
  * Presence of antimitochondrial antibody (immunofluorescence titer ≥ 1:40 or positive antigen-specific test), specific antinuclear immunofluorescence (nuclear dots or perinuclear rims) or positive antigen-specific test for anti-gp210 or anti-Sp100 antibodies
  * Records of histologic features suggestive of, or compatible with PBC
* UDCA therapy for the past 12 months (stable dose ≥ 12 mg/kg/d for ≥ 3 months prior to inclusion).
* Non-optimal response to UDCA defined by at least one of the following criteria (ratios of absolute values to ULN rounded to the first decimal digit) observed at least 2 times at ≥ 4 weeks interval in the past 3 months, including at the inclusion visit assessment:
* ALP > 1.0 xULN
* GGT > 3.0 xULN
* ALT or AST > 1.0 xULN
* Total and conjugated bilirubin > 1.0 xULN
* Women of childbearing potential must use at least one barrier contraceptive during the study and for at least 90 days after the last dose.
* Affiliation to a social security system (AME excepted).
* Signed informed consent.

Exclusion Criteria:

* Any of the following signs of advanced chronic liver disease:

  * Total bilirubin > 2.0 xULN
  * Serum albumin < 32 g/l
  * Platelet count < 100,000/mm3
  * INR > 1.3 or prothrombin index < 60%
  * Child-Pugh score B or C
  * MELD score ≥ 14
  * History ≤ 24 months or presence of cirrhotic decompensation
  * Patients on the waiting list for LT
* GFR estimated by CKI-EPI equation < 60 mL/min
* CPK > 5.0 xULN
* AST or ALT > 3.0 xULN
* History of LT
* Autoimmune hepatitis (AIH) overlap syndrome defined by at least 2 of the following 3 criteria including the histologic one:

  * ALT > 5.0 xULN
  * IgG > 20 g/l or presence of anti-smooth muscle or anti-SLA antibodies
  * Histologic features characteristic of, or compatible with AIH
* Any other chronic hepatic comorbidities (HCV, HBV, NASH, alcoholic liver disease, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, celiac disease)
* Untreated hypo or hyperthyroidism (Hashimoto or Graves autoimmune thyroiditis)
* Conditions that may cause non-hepatic increases in ALP (Paget's disease, osteodystrophy, hyperparathyroidism, dysglobulinemia)
* Gilbert's syndrome or chronic hemolysis (hyperbilirubinemia with an unconjugated to total bilirubin ratio ≥ 75%)
* History of or established or suspected hepatocellular carcinoma
* History of malignancy diagnosed or treated within 2 years (recent localized treatment of squamous or non-invasive basal skin cancers is permitted)
* Any severe comorbidity that may reduce life expectancy ≤ 2 years
* Pregnancy or lactating
* Known intolerance to bezafibrate
* Known hypersensitivity to bezafibrate, any of the components of Befizal© or other fibrates
* Known photosensitivity reactions or photoallergy reactions to fibrates
* Patient with congenital galactosemia, glucose malabsorption, or lactase deficiency because of presence of lactose in LP tablets of bezafibrate
* Participation in any other interventional study in the past 6 months
* Any of the following medications used in the past 3 months before inclusion: bezafibrate, fenofibrate, ciprofibrate, gemfibrozil, obeticholic acid, budesonide, any other systemic corticosteroids, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus, sirolimus, everolimus, methotrexate.
* Use of statins in the month before inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of bezafibrate 200 mg and bezafibrate 400 mg versus placebo as adjunctive treatments in patients with PBC and a non-optimal response to UDCA. | Week 48
  Proportion of patients with a complete biochemical response defined by normal serum levels of alkaline phosphatase (ALP), gamma-glutamyl transpeptidase (GGT), aminotransferases (AST, ALT), and total bilirubin at 48 weeks of treatment.

SECONDARY OUTCOMES:
To compare adverse effects between groups, in particular on muscle, kidney, and liver. | Week 48 and Week 96 ( extension phase)
  Proportion of patients with serious adverse events (SAE) and/or adverse events (AE) at W48 and W96 (extension phase), including creatinine > 150 μmol/L, CPK > 10 xULN, or ALT > 5 xULN.
To compare symptoms (Pruritus) between groups | Week 48 and Week 96 (extension phase)
  Proportion of patients with significant pruritus based on worst itch numerical rating scale (WI-NRS).
To compare symptoms (fatigue) between groups. | Week 48 and Week 96 (extension phase)
  Proportion of patients with significant fatigue at W48 and W96 based on PBC-40 questionnaire.
To compare quality of life (QoL) between groups. | Week 48 and Week 96 (extension phase)
  Changes from baseline to W48 and W96 in quality of life assessed by PBC-40.
Level of liver biochemical parameters between groups | Week 48 and Week 96 (extension phase)
  Proportion of patients with a deep biochemical response defined by normal levels of ALP, GGT, ALT, AST, and a total bilirubin ≤ 0.6 mg/dL.
Changes in liver stiffness by Fibroscan | Week 48 and Week 96 (extension phase)
  To compare changes in non-invasive markers of liver fibrosis between groups.
Changes in liver stiffness (Fibroscan) by ELF test. | Week 48 and Week 96 (extension phase)
  To compare changes in non-invasive markers of liver fibrosis between groups.
Changes in liver stiffness (Fibroscan) by FIB-4 score. | Week 48 and Week 96 (extension phase)
  To compare changes in non-invasive markers of liver fibrosis between groups.
Proportion of patients with advanced fibrosis or cirrhosis as diagnosed by Fibroscan | Week 48 and Week 96 (extension phase)
  To compare changes in non-invasive markers of liver fibrosis between groups.
Proportion of patients with moderately advanced or advanced disease as diagnosed by the Rotterdam criteria | Week 48 and Week 96 (extension phase)
  To compare changes in non-invasive markers of liver fibrosis between groups.
To compare occurrence of clinical events including death, LT, or liver complications between groups. | Week 48 and Week 96 (extension phase)
  Occurrence of all-cause and liver-related deaths, LT, referral for LT, ascites, spontaneous bacterial peritonitis, variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, hepatocellular carcinoma, unscheduled hospitalization, development of any new comorbidities or significant worsening of preexisting ones at W48 and W96.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Corpechot, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hepatology department - Hospital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No